CLINICAL TRIAL: NCT02409953
Title: Effect of Immersion, Performed Under the Conditions of Obstetrical Dilatation Bath, on Diuresis and Hemodynamic Variables in Young Women
Acronym: IMMERSION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5979
Record Dates: First submitted 2015-03-24; First posted 2015-04-07 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Healthy
Keywords: volunteers
MeSH Terms: interventions — Supine Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bath (Experimental)
  Interventions: Other: Lying in a bath during 2 hours
- Bed (Placebo Comparator)
  Interventions: Other: Lying in a bed during 2 hours

INTERVENTIONS:
Other: Lying in a bath during 2 hours
  Arms: Bath
Other: Lying in a bed during 2 hours
  Arms: Bed

SUMMARY:
Like in the full immersion, studied in the context of diving, immersion in water causes a cascade of events with hemodynamic and hormonal consequences.

First, immersion leads to a relative hypervolemia by venous redistribution and then 40-60 minutes later, hypovolemia by stimulating diuresis.

Dilatation bath is helpful in relieving moderate pain the first stage of obstetrical labor.

However, when the labor progresses, the dilatation bath is no longer sufficient and epidural analgesia remains the only effective method to control pain.

Used before the realization of an epidural analgesia, dilatation bath could affect blood volume and thus worsen the hemodynamic consequences of the sympathetic block that is linked to the installation of sensory block of the epidural analgesia in the parturient (severe prolonged maternal hypotension that can cause a decrease of the placental perfusion and fetal distress).

Before beginning a study in pregnant women, it seems essential to study the hemodynamic consequences of the dilatation bath in a comparable population of volunteers healthy young women and out of the obstetrical context.

ELIGIBILITY:
Inclusion Criteria:

Healthy female volunteers aged 18 to 45 years

Exclusion Criteria:

* pregnancy
* menopause (confirmed for at least 12 weeks)
* breastfeeding
* Proteinuria> 2 cross on the dipstick
* Glycosuria > 2 cross on the dipstick
* subject with no empty stomach for at least 8 hours
* Taking medication in the week before the test affecting diuresis, production of antidiuretic hormone or on the cardiovascular system: paracetamol, nonsteroidal anti-inflammatory Alcohol intake the day before the tes

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04-15; Primary Completion 2016-05-13 (Actual); Study Completion 2016-05-13 (Actual)

PRIMARY OUTCOMES:
diuresis (urine volume in milliliters) | 120 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie - Réanimation Chirurgicale de Hautepierre, Strasbourg, Alsace, France

IPD SHARING:
Plan to Share IPD: No